CLINICAL TRIAL: NCT05359913
Title: Proof of Concept and Feasibility in Podcasting Cervical Cancer Prevention for African American Women
Brief Title: Podcasting Cervical Cancer Prevention for AAW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Chakema Carmack, Associate Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003472
Record Dates: First submitted 2022-04-07; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; African American Women; Cancer Prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- African American Women (Experimental)
  Interventions: Behavioral: Cervical cancer podcast for African American women

INTERVENTIONS:
Behavioral: Cervical cancer podcast for African American women — The video podcast will deliver cervical cancer prevention messages using entertainment education and behavioral journalism, and film production techniques such as "talking head" video, interview, animations, & live-action skits. The research team will work closely with the production company in scripting the video vignettes and sequences, ensuring that video content reflects salient domains captured in the concept mapping research development phase of the study.

SUMMARY:
For African American women (AAW) in Houston, cervical cancer mortality is disproportionate to their racial and ethnic counterparts.Most notably, lack of human papillomavirus (HPV) screening, vaccination, and later diagnosis increase cervical cancer mortality. However, cervical cancer is largely preventable. While previous research has identified only a few social determinants that are specifically related to cervical cancer, there may be a host of additional social and cultural factors that contribute to a lack of preventative behavior. The overall objective of the proposed study is to gather preliminary data to determine whether the use of concept mapping methodology is useful in identifying unique sociocultural determinants of cervical cancer prevention behavior, and to pilot test the feasibility of a podcast video developed using the information garnered from the concept mapping procedure. It is hypothesized that the resulting podcast video will increase HPV knowledge and behavioral intentions. Proof of concept and feasibility are needed first, in determining the utility of both the methodology and media development procedures, as well as data on preliminary effect outcomes, before further investigation and program development.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as African American
* biological female sex
* speak and read English
* 18 years old or older
* not currently or previously diagnosed with cervical cancer or cervix dysplasia

Exclusion Criteria:

• history of hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Researcher-developed cervical cancer prevention measure that reflects salient socio-cultural perceptions of cervical cancer prevention (obtained through non-clinical qualitative inquiry) | To be measured immediately before film viewing and immediately after film viewing
  To observe whether the podcast video significantly changed perceptions of cervical cancer prevention.
  Items will be set to 5-pt Likert-type scale: (1) - (5); higher scale values indicating more positive perceptions to cervical cancer prevention
Pap test intentions: Do you intend to obtain a Pap cytology screening? (single item) | To be measured immediately before film viewing and immediately after film viewing
  To observe whether the podcast video significantly changed intentions to obtain a Pap cytology test.
  Item will be set to 5-pt Likert-type scale: (1) - (5); higher scale values indicating greater intentions for cervical cancer screening.
HPV vaccination intentions: Do you intend to get vaccinated for HPV? (single item) | To be measured immediately before film viewing and immediately after film viewing
  For women who are within the HPV vaccination age range: to observe whether the podcast video significantly changed their intentions to obtain a HPV vaccination.
  Items will be set to 5-pt Likert-type scale: (1) - (5); higher scale values indicating more positive intentions toward HPV vaccination.

IPD SHARING:
Plan to Share IPD: No
Because this is a feasibility study with a very low sample size, the data is preliminary and it is not certain that the data will be appropriate or useful for public dissemination.